CLINICAL TRIAL: NCT01111994
Title: Efficacy & Safety of Clindamycin Phosphase 1.2% and Tretinoin 0.025% Gel vs. Vehicle for the Treatment of Acne and Acne-Induced Post Inflammatory Hyperpigmentation in Patients With Skin of Color
Brief Title: Efficacy & Safety of Clindamycin and Tretinoin in Acne
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Callender Center for Clinical Research (Other)
Collaborators: Society Hill Dermatology (Other)
Responsible Party: Valerie D. Callender, M.D., Callender Center for Clinical Research
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: VDC2009Z
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-05

CONDITIONS: Acne
Keywords: hyperpigmentation
MeSH Terms: conditions — Acne Vulgaris; Hyperpigmentation | interventions — clindamycin phosphate; Tretinoin; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clindamycin Phosphate 1.2% and Tretinoin 0.025% Gel — Clindamycin Phosphate 1.2% and Tretinoin 0.025% Gel QD for 3 months
  Other Names: Ziana Gel

SUMMARY:
The purpose of this study is ascertain the efficacy and safety of Clindamycin

Phosphate 1.2% and Tretinoin 0.025% in the treatment of Acne and Post

Inflammatory Hyperpigmentation in patients with skin of color.

DETAILED DESCRIPTION:
Acne is a chronic disorder of the pilosebaceous glands characterized by

inflammatory papules, pustules, opened and closed comedones, cysts and

nodules. Post inflammatory hyperpigmentation is a condition in which an

inflammation from a disease such as acne, trauma, or abrasion results in areas

of the skin with increased melanin content compared to the surrounding skin.

There are several treatments available for acne, which include benzoyl

peroxide,antibiotics (topical or oral), and topical retinoids (tretinoin,

tazarotene, adapalene). Combination therapy, such as topical retinoid and

clindamycin, has been shown to be more effective than monotherapy in

addressing all pathogenic factors of acne.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate facial acne and mild to moderate post-inflammatory hyperpigmentation
* Photo skin types IV - VI
* Ages 12 and older
* Both sexes
* Two week washout period for topical anti-acne medications, medicated cosmetics,and bleaching products
* Thirty day washout period for oral corticosteroids, oral antibiotics,and oral contraceptives

Exclusion Criteria:

* Seborrheic dermatitis
* PIH of solely dermal origin
* Acne vulfaris known to be resistant to oral antibiotics
* Use of erythromycin-containing products
* Use of neuromuscular blocking agents
* Pregnancy, breastfeeding, a positive pregnancy test in the office, or plans to become pregnant. Women of childbearing age must use reliable forms of contraception (e.g., abstinence, oral contraceptives, or spermicide and condoms).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Improvement of acne and post inflammatory hyperpigmentation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Callender, MD, Principal Investigator — Callender Center for Clinical Research
Locations (2):
- United States (2):
  - Callender Center for Clinical Research, Mitchellville, Maryland
  - Society Hill Dermatology, Philadelphia, Pennsylvania